CLINICAL TRIAL: NCT00355004
Title: Improving Systems for Colorectal Cancer Screening
Brief Title: Computerized and Mailed Reminders in Increasing the Rate of Colorectal Cancer Screening in Adults With an Average Risk for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Screening
Other Study IDs: CDR0000486405; HMS-M11960-103; HCHP-1305
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-01

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling; Occult Blood

INTERVENTIONS:
Other: counseling intervention
Procedure: fecal occult blood test
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Screening may help doctors find colorectal cancer sooner, when it may be easier to treat. Computerized and mailed reminders may help increase the rate of colorectal cancer screening in adults with an average risk for colorectal cancer.

PURPOSE: This randomized clinical trial is studying how well computerized and mailed reminders work in increasing the rate of colorectal cancer screening in adults with an average risk for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether rates of colorectal cancer (CRC) screening can be increased among average-risk adults by using patient-specific, active, electronic, clinical reminders for primary care physicians during office visits and mailed reminders and fecal occult blood test cards for patients.

Secondary

* Calculate baseline rates of CRC screening, in terms of patient demographic characteristics, primary care physician, and practice group, by using computerized clinical information systems to identify patients due for screening.
* Assess baseline rates of CRC screening among patients insured by different health plans.
* Determine whether the impact of the interventions is related to efforts by health plans to promote CRC screening.
* Evaluate patients' willingness to use a validated web-based tool to estimate their personal risk of CRC.

OUTLINE: This is a randomized, controlled study. Patients are randomized to 1 of 2 arms (arms I or III). Physicians are randomized to 1 of 2 arms (arms II or IV).

* Arm I: Patients receive mailed reminders for colorectal cancer (CRC) screening. Patients also receive fecal occult blood testing (FOBT) instructions and cards. Patients who remain overdue for screening at 6 months after the initial mailing receive a follow-up letter reminding them of their need to be screened. Patients who return positive FOBT cards undergo colonoscopy within 1 month. The patient's primary care physician may receive computerized screening reminders at the time of the patient's office visit and may order CRC screening tests online.
* Arm II: Patients receive no mailings. The patient's primary care physician may receive computerized screening reminders at the time of the patient's office visit and may order CRC screening tests online.
* Arm III: Patients receive mailed reminders for CRC screening. The patient's primary care physician may order CRC screening tests online, but will not receive active computerized reminders. Patients also receive FOBT instructions and cards. Patients who remain overdue for screening at 6 months after the initial mailing receive a follow-up letter reminding them of their need to be screened. Patients who return positive FOBT cards will be scheduled to undergo colonoscopy within 1 month.
* Arm IV: Patients receive no mailings. The patient's primary care physician may order CRC screening tests online, but will not receive active computerized reminders.

Patients are followed for 15 months to determine screening rates.

PROJECTED ACCRUAL: A total of 21,860 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Receiving primary care at 1 of 11 participating Harvard Vanguard Medical Associates (HVMA) centers

  * Has an active primary care physician
  * Had a primary care visit within the past 18 months
* Is due for colorectal cancer screening

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21860 (Estimated)
Dates: Start 2005-03; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Rate of colorectal cancer screening

SECONDARY OUTCOMES:
Number of patients with adenomatous polyps and colon cancer diagnosed
Number of stool cards returned and abnormal stool cards
Number and dates of sigmoidoscopies and colonoscopies scheduled and performed

CONTACTS AND LOCATIONS:
Overall Officials: John Ayanian, MD, MPP, Study Chair — Harvard Medical School (HMS and HSDM); Robert H. Fletcher, MD — Harvard Pilgrim Health Care
Locations (3):
- United States (3):
  - Harvard Medical School, Boston, Massachusetts
  - Harvard Pilgrim Health Care, Boston, Massachusetts
  - Harvard Vanguard Medical Associates - Kenmore, Boston, Massachusetts

REFERENCES:
- [Result] Sequist TD, Zaslavsky AM, Marshall R, Fletcher RH, Ayanian JZ. Patient and physician reminders to promote colorectal cancer screening: a randomized controlled trial. Arch Intern Med. 2009 Feb 23;169(4):364-71. doi: 10.1001/archinternmed.2008.564. PMID 19237720